CLINICAL TRIAL: NCT01722669
Title: Pharmacokinetic and Pharmacodynamic Study of Oral Quercetin and Isoquercetin in Healthy Adults and Patients With Hypercoagulable States.
Brief Title: Quercetin PK/PD Study in Healthy Adults and Patients With Hypercoagulable States
Acronym: PK/PD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jeff Zwicker, Associate Professor, Harvard Medical School, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012P000022
Record Dates: First submitted 2012-05-10; First posted 2012-11-07 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Healthy
Keywords: quercetin; isoquercetin; pharmacokinetic; pharmacodynamic
MeSH Terms: interventions — isoquercitrin; Quercetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Quercetin (Experimental): Single dose of quercetin with or without ascorbic acid
  Interventions: Drug: isoquercetin or quercetin
- Isoquercetin (Active Comparator): Single dose of isoquercetin with or without ascorbic acid
  Interventions: Drug: isoquercetin or quercetin

INTERVENTIONS:
Drug: isoquercetin or quercetin — Single dose PK/PD study

SUMMARY:
The goal of this study is to evaluate how much quercetin or isoquercetin is absorbed after a single dose and evaluate for pharmacokinetic inhibition of protein disulfide isomerase. Pharmacodynamic studies will also be performed in an additional cohort of 10 patients with evidence of antiphospholipid antibodies

DETAILED DESCRIPTION:
To compare the absorption and activity of quercetin or isoquercetin with or without ascorbic acid in healthy adults. Oral chews containing quercetin (500mg) or isoquercetin(500 mg total) with or without ascorbic acid will be given. Pharmacokinetic parameters (AUC, Cmax, Tmax, elimination half-life) will be determined over 24 hours (8 time points). Pharmacodynamic inhibition of protein disulfide isomerase activity will also be assessed.

In addition to healthy subjects, a cohort of 10 individuals with antiphospholipid antibodies will participate. These participants will receive isoquercetin 1000 mg and have pharmacodynamics studies performed at time 0 and 4 hours.

All study drugs will be provided by Quercegen Pharma.

ELIGIBILITY:
Inclusion Criteria

* Subject is willing to participate and provide informed consent
* Subject is considered reliable and capable of adhering to the protocol per the judgment of the Investigator
* Subjects in group D must exhibit good organ reserves (within prior 4 weeks) defined as:

  1. Estimated GFR >35 (formula),
  2. Platelet count >65 K/uL,
  3. Hemoglobin >10.5 grams/dL
  4. Total bilirubin <2.0 mg/dL
* Minimum age 18 years old
* Body mass index (BMI) between 18 and 35 kg/m2
* For cohort D (antiphospholipid antibodies) a. Subjects in group D must have at least one positive antiphospholipid antibody within the last 8 weeks and/or previous confirmed antibodies (2 or more occasions at least 12 weeks apart) : i. Positive lupus anticoagulant ii. anticardiolipin antibody IgM or IgG (>40U GPL) iii. anti-β2 Glycoprotein1 antibody titer (>35 units)

Exclusion Criteria

* Pregnant. If female of child-bearing age, negative urinary pregnancy test prior to dosing of quercetin or isoquercetin
* No history of malabsorptive gastrointestinal disorder
* Currently taking aspirin, NSAIDS, warfarin, low-molecular weight heparin or other anticoagulants (such as direct thrombin inhibitors or factor X inhibitors)

  a. Note: Study subjects taking aspirin or NSAIDS, if treating physician concurs, are permitted to enroll if plan to hold for aspirin 10 days or NSAIDS 24 hours prior to dosing of quercetin/isoquercetin
* Prescribed niacin for hyperlipidemia
* Known HIV
* History of sensitivity or intolerance to flavonoids, niacin or ascorbic acid
* May not have uncontrolled intercurrent illness including, but not limited to ongoing or active infection, hepatitis, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-05; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zwicker, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Contact PI
Supporting Information: Study Protocol
Time Frame: 3 years

REFERENCES:
- [Derived] Stopa JD, Neuberg D, Puligandla M, Furie B, Flaumenhaft R, Zwicker JI. Protein disulfide isomerase inhibition blocks thrombin generation in humans by interfering with platelet factor V activation. JCI Insight. 2017 Jan 12;2(1):e89373. doi: 10.1172/jci.insight.89373. PMID 28097231

RESULTS

PARTICIPANT FLOW:
Groups:
- Quercetin 500mg (ARM A1): Single dose PK/PD analyses of quercetin 500 mg
- Isoquercetin 500mg (ARM B1): Single dose PK/PD of isoquercetin 500 mg
- Quercetin 500 mg + Ascorbic Acid (ARM A2): Single dose quercetin with 500 mg + ascorbic acid pk/pd analyses
- Isoquercetin 500 mg + Ascorbic Acid (ARM B2): Single dose isoquercetin 500 mg + ascorbic acid pk/pd analyses
- Isoquercetin 1000 mg + Ascorbic Acid (ARM C): Single dose isoquercetin + 1000 mg ascorbic acid
- Antiphospholipid Antibody Cohort (ARM D): Single dose isoquercetin 1000 mg + 1000 mg ascorbic acid in patients with antiphospholipid antibodies
Period: Overall Study
Arm/Group | Quercetin 500mg (ARM A1) | Isoquercetin 500mg (ARM B1) | Quercetin 500 mg + Ascorbic Acid (ARM A2) | Isoquercetin 500 mg + Ascorbic Acid (ARM B2) | Isoquercetin 1000 mg + Ascorbic Acid (ARM C) | Antiphospholipid Antibody Cohort (ARM D)
Started | 5 | 5 | 5 | 5 | 10 | 8 (Antiphospholipid Antibody (ARM D): 6 evaluable and 2 withdrew consent without any data collected)
Completed | 5 | 5 | 5 | 5 | 10 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Measure Analysis Population Description: Antiphospholipid Antibody (ARM D): 2 withdrew consent without any data collected
Groups:
- Quercetin 500 mg (ARM A1): Single dose of quercetin PK/PD analysis
- Isoquercetin 500 mg (ARM B1): Single dose of isoquercetin PK/PD analysis
- Quercetin 500 mg + Ascorbic Acid (ARM A2): Single dose of quercetin + ascorbic acid PK/PD analysis
- Isoquercetin 500 mg + Ascorbic Acid (ARM B2): Single dose of isqouercetin +ascorbic acid PK/PD analysis
- Isoquercetin 1000 mg + Ascorbic Acid (ARM C): single dose isoquercetin + ascorbic acid PK/PD analyses
- Antiphospholipid Antibody (ARM D): single dose isoquercetin +ascorbic acid in patients with antiphospholipid antibodies
- Total: Total of all reporting groups
Arm/Group | Quercetin 500 mg (ARM A1) | Isoquercetin 500 mg (ARM B1) | Quercetin 500 mg + Ascorbic Acid (ARM A2) | Isoquercetin 500 mg + Ascorbic Acid (ARM B2) | Isoquercetin 1000 mg + Ascorbic Acid (ARM C) | Antiphospholipid Antibody (ARM D) | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 10 | 6 | 36
Age, Categorical [Count of Participants; unit: Participants] — Population: Antiphospholipid Antibody (ARM D): 2 withdrew consent without data collected
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 5 | 5 | 5 | 5 | 10 | 4 | 34
    >=65 years | 0 | 0 | 0 | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Antiphospholipid Antibody (ARM D): 2 withdrew consent without data collected
  Participants
    Female | 2 | 3 | 2 | 3 | 5 | 5 | 20
    Male | 3 | 2 | 3 | 2 | 5 | 1 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Antiphospholipid Antibody (ARM D): 2 withdrew consent without data collected
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 0 | 2
    Not Hispanic or Latino | 2 | 1 | 2 | 1 | 5 | 6 | 17
    Unknown or Not Reported | 3 | 4 | 3 | 4 | 3 | 0 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Antiphospholipid Antibody (ARM D): 2 withdrew consent without data collected
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 1 | 1 | 1 | 1 | 1 | 0 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 1 | 0 | 1 | 0 | 0 | 1 | 3
    White | 2 | 2 | 2 | 2 | 5 | 5 | 18
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 2 | 1 | 2 | 4 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: AUC 0-24 hours of measured plasma quercetin aglycone for Arms A1, B1, A2, B2, C Collected at timepoints: baseline and 1, 2, 4, 6, 8, and 24 hours after dose. PK and PDI samples were not measured for Arm D (anti-phospholipid antibody cohort)
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: uM hr/L
Groups:
- Quercetin 500 mg (ARM A1); Isoquercetin 500 mg (ARM B1); Quercetin 500 mg + Ascorbic Acid (ARM A2); Isoquercetin 500 mg + Ascorbic Acid (ARM B2); Isoquercetin 1000 mg + Ascorbic Acid (ARM C): Single dose, measurement of plasma quercetin aglycone
Arm/Group | Quercetin 500 mg (ARM A1) | Isoquercetin 500 mg (ARM B1) | Quercetin 500 mg + Ascorbic Acid (ARM A2) | Isoquercetin 500 mg + Ascorbic Acid (ARM B2) | Isoquercetin 1000 mg + Ascorbic Acid (ARM C)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 10
uM hr/L | 4.78 (1.67) | 15.00 (8.94) | 5.41 (2.13) | 16.34 (10.08) | 40.3 (17.11)

2. Secondary Outcome: Reductase Activity of PDI Using Dieosin Glutathione Disulfide
Description: Measurement of protein disulfide inhibition in plasma using a fluorescent PDI substrate (dieosin glutathione disulfide)
Time Frame: 2 hours. Not measured in D
Population: 2 hours after oral ingestion
Measure: Mean (Standard Deviation); unit: Percent inhibition
Groups:
- Quercetin 500 mg (ARM A1); Isoquercetin 500 mg (ARM B1); Quercetin 500 mg + Ascorbic Acid (ARM A2); Isoquercetin 500 mg + Ascorbic Acid (ARM B2); Isoquercetin 1000 mg + Ascorbic Acid (ARM C): PDI activity measured by DiESSG assay at 0 and 2 hours
Arm/Group | Quercetin 500 mg (ARM A1) | Isoquercetin 500 mg (ARM B1) | Quercetin 500 mg + Ascorbic Acid (ARM A2) | Isoquercetin 500 mg + Ascorbic Acid (ARM B2) | Isoquercetin 1000 mg + Ascorbic Acid (ARM C)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 10
Percent inhibition | 31.9 (24.14) | 63.2 (25.3) | 16 (31.8) | 8.3 (15.03) | 38 (35)

3. Secondary Outcome: Platelet-induced Thrombin Generation (U/mL)
Description: Thrombin induced thrombin generation measured in patient plasma
Time Frame: 4 hours
Population: 4 hours after single dose only measured in Arm C and Arm D
Measure: Mean (Standard Deviation); unit: U/mL
Groups:
- Isoquercetin 1000 mg + Ascorbic Acid (ARM C): Thrombin induced thrombin generation measured before and after isoquercetin + Ascorbic acid at time 0 and 4 hours
- Antiphospholipid Antibody (ARM D): Thrombin induced thrombin generation measured at time 0 and 4 hours following isoquercetin 1000 mg
Arm/Group | Isoquercetin 1000 mg + Ascorbic Acid (ARM C) | Antiphospholipid Antibody (ARM D)
Number analyzed (Participants) | 10 | 6
U/mL | 0.30 (.28) | 1.40 (2.14)

ADVERSE EVENTS:
Time Frame: Assessed during visit 1, up to 24 hours
Groups:
- Quercetin 500 mg (ARM A1); Isoquercetin 500 mg (ARM B1): Toxicity over 24 hours following single dose
- Quercetin 500 mg + Ascorbic Acid (ARM A2): Toxicity over 24 hours following single dose of combined quercetin and ascorbic acid
- Isoquercetin 500 mg + Ascorbic Acid (ARM B2): Toxicity over 24 hours following single dose of combined isoquercetin and ascorbic acid
- Isoquercetin 1000 mg + Ascorbic Acid (ARM C); Antiphospholipid Antibody (ARM D): Toxicity over 24 hours following single dose of isoquercetin
Arm/Group | Quercetin 500 mg (ARM A1) | Isoquercetin 500 mg (ARM B1) | Quercetin 500 mg + Ascorbic Acid (ARM A2) | Isoquercetin 500 mg + Ascorbic Acid (ARM B2) | Isoquercetin 1000 mg + Ascorbic Acid (ARM C) | Antiphospholipid Antibody (ARM D)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/10 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT01722669/Prot_SAP_000.pdf